CLINICAL TRIAL: NCT06868602
Title: Effects of Regular Exercise and Psychoeducation on Quality of Life, Depression and Physical Function in the Treatment of Sarcopenia in Elderly Individuals
Brief Title: Effects of Regular Exercise and Psychoeducation on Quality of Life and Depression in the Treatment of Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Elif Asan, clinical physiotherapist, Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-664; BAP01-2024-5152 (Other Grant/Funding Number: Ondokuz Mayıs University)
Record Dates: First submitted 2025-02-25; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Sarcopenia in Elderly
Keywords: sarcopenia; exercise; psychoeducation
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: In this study, a pre-test-post-test randomized control and placebo group quasi-experimental research design will be used.
  In order to determine whether elderly individuals who voluntarily accept to participate in the study are sarcopenic according to the definitive diagnostic criteria of the European Working Group (EWGSOP2), muscle strength assessment (with a handheld dynamometer), muscle mass assessment (with a Bioelectrical Impedance (BIA) device) and Physical performance assessment (with the Timed Up and Go test and SARC-F test) will be performed; then, the SMMT will be applied to sarcopenic individuals and those who score 24 points and above and meet the inclusion criteria will be included in the study.
  Elderly individuals who meet the inclusion criteria will be assigned to the group where exercise will be performed, the group where exercise and psychoeducation will be done together, and the control group.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention): This group will be informed about exercise and psychoeducation only once after the sessions are completed.
- exercise (Active Comparator): Physical exercise will be performed for 45 minutes twice a week for eight weeks.
  Interventions: Other: Exercise
- exercise and psychoeducation (Active Comparator): A 45-minute exercise program twice a week and a 45-minute psychoeducation program once a week will be implemented for 8 weeks.
  Interventions: Other: psychoeducation; Other: Exercise

INTERVENTIONS:
Other: psychoeducation — Although the literature investigating the effectiveness of exercise programs on quality of life, physical function and depression in sarcopenic individuals is extensive, no studies have been found in which psychoeducation programs are applied to sarcopenic individuals and their effectiveness is investigated. In this planned study,Researchers aim to observe what kind of results will emerge and in what direction the psychoeducation program will shape the treatment by applying both exercise and psychoeducation programs to sarcopenic individuals.
  Other Names: exercise
  Arms: exercise and psychoeducation
Other: Exercise — Although the literature investigating the effectiveness of exercise programs on quality of life, physical function and depression in sarcopenic individuals is extensive, no studies have been found in which psychoeducation programs are applied to sarcopenic individuals and their effectiveness is investigated. In this planned study, Researchers aim to observe what kind of results will emerge and in what direction the psychoeducation program will shape the treatment by applying both exercise and psychoeducation programs to sarcopenic individuals.
  Arms: exercise; exercise and psychoeducation

SUMMARY:
In this study, it was aimed to observe the effect of psychoeducation, which has not yet been included among the treatment methods of sarcopenia, which affects elderly individuals both physically and psychologically and has been proven to negatively affect their quality of life, on Quality of Life, Depression and Physical Function when applied with exercise therapy.

It is known that exercise programs applied in the treatment of sarcopenia, which has become a common problem in elderly individuals and is known as the trigger of most symptomatic diseases, have positive effects.

However, no psychoeducation program has been applied to date in the treatment of sarcopenia, which is thought to trigger psychological factors as well as physical factors.

In this direction, it is aimed to contribute to sarcopenia treatment and indirectly to geriatric rehabilitation programs according to the results we will obtain in sarcopenic individuals with the psychoeducation program, which we think is lacking.

In addition to all these, sarcopenia, which is a treatable diagnosis and one of the biggest obstacles to the independent life of elderly individuals, is thought to be a preventable condition with preventive rehabilitation programs.

Researchers believe that preventive rehabilitation programs will positively affect the amount spent on elderly care services, which constitute a large portion of our country's health expenses, and Researchers aim to support these issues with the results they will obtain.

DETAILED DESCRIPTION:
This study was planned to examine the effectiveness of exercise and psychoeducation programs applied to sarcopenic individuals.

Sarcopenia, which causes muscle strength loss in elderly individuals, is shown as a risk factor for many negative outcomes ranging from fractures to death.

Sarcopenia, which is also shown as the cause of many metabolic diseases, is often a preventable disease, but it is seen that scientific studies on sarcopenia treatment in the academic field are not sufficient.

While the majority of the studies conducted include physiotherapy programs, the psychological dimension of the treatment has been ignored and although it has been associated with depression, no scientific study has been found that includes this psychoeducation program.

The physical problems experienced by sarcopenic individuals are basically movement disorders that occur due to muscle strength loss, along with deterioration in their quality of life and physical functions, and musculoskeletal system diseases.

However, sarcopenia is a multifaceted disease that is not only physical but also causes psychological diseases such as depression.

In addition, it is known that physical function loss, which is one of the symptoms of sarcopenia, has a negative effect on the level of depression, independent of sarcopenia.

In light of all this information, it is thought that if the treatment program prepared for sarcopenic individuals does not include a psychoeducation program together with the physiotherapy program, a part of the treatment will be incomplete.

This study, which researchers designed to investigate the psychoeducation program, the therapeutic effect of which is not yet known on sarcopenia, aims to contribute to this area.

It is aimed to reach a conclusion by comparing the differences between the Physical Function, Quality of Life and Depression parameters of the psychoeducation program combined with the exercise program in sarcopenic individuals and the sarcopenic individuals who only received the exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 60 and over who have signed a consent form and agreed to volunteer for the study.
* Individuals classified as sarcopenic according to the criteria of the European Working Group on Sarcopenia (EWGSOP2).
* Individuals who scored 24 points or higher on the Standardized Mini Mental Test.

Exclusion Criteria:

* Individuals with neurological disease,
* Individuals with advanced kidney disease,
* Individuals with pacemakers,
* Individuals with advanced vision and hearing problems,
* Individuals with advanced dementia,
* Individuals with orthopedic disabilities

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
TUG test | Before treatment
  A chair and a stopwatch are required for the test, which evaluates the risk of falls and mobility in the elderly. The test is performed with the shoes the individual always uses. A 3-meter area is determined in front of the chair. The individual is asked to get up from the chair, walk this distance, and sit down again.
SF-12 Test | Before treatment
  It is an abbreviated form for assessing quality of life. This form, developed by Ware et al. (1995), is not specific to any age or type of disease, but is a scale that assesses the person's quality of life over the last four weeks. SF-12; It includes the sub-elements of physical functioning, physical role, pain, general health, emotional role, mental health, social functioning and vitality and consists of 12 questions.
GDS | Before treatment
  This scale was developed by Yesavage et al. (1983). The Turkish adaptation of the scale was made by Ertan et al. The scale is self-reporting, aimed at the elderly, easy to answer and consists of 30 questions. A higher score indicates a higher level of depression.
Bioelectrical impedance analysis (BIA) | Before treatment
  Bioelectrical impedance analysis (BIA) measurement; It is a non-invasive measurement. It takes advantage of the different resistance of different tissues in the body to currents. A weak electric current is directed to the body and the impedance is measured. It is used to estimate body composition parameters such as total body water and fat-free mass.
SARC-F | Before treatment
  SARC-F; It allows health professionals to quickly and easily assess the risk of sarcopenia in primary health care. It asks 5 questions about "strength, assistance while walking, getting up from a chair, climbing stairs and falling". The SARC-F score range is from 0 to 10, with a score range of 0-3 representing a healthy condition and a score range of 4 and above representing a symptomatic condition.
Standardized Mini Mental Test (SMMT) | Before treatment , pre test only
  Mini Mental Test developed by Folstein et al. (1975) allows for cognitive assessment in a short time. In this respect, SMMT is a short, easy-to-apply and standardized test used to determine the cognitive level globally.
Handgrip strength assessment | Before treatment
  During the assessment, the individual is seated upright on a chair without surface support for the arm being assessed. The arm to be measured is positioned in a free position, with the knee angle and elbow angle at 90 degrees. The subject is asked to squeeze the dynamometer with their fingers as hard and tight as possible. The measurements are repeated 3 times, with 10 seconds between them and each measurement being no less than 5 seconds, and any interventions that may affect the measurements during the assessment are avoided.

SECONDARY OUTCOMES:
TUG test | Within a week of the end of treatment (within 1 week of the completion of the 8-week treatment)
  A chair and a stopwatch are required for the test, which evaluates the risk of falls and mobility in the elderly. The test is performed with the shoes the individual always uses. A 3-meter area is determined in front of the chair. The individual is asked to get up from the chair, walk this distance, and sit down again.
SF-12 Test | Within a week of the end of treatment (within 1 week of the completion of the 8-week treatment)
  It is an abbreviated form for assessing quality of life. This form, developed by Ware et al. (1995), is not specific to any age or type of disease, but is a scale that assesses the person's quality of life over the last four weeks. SF-12; It includes the sub-elements of physical functioning, physical role, pain, general health, emotional role, mental health, social functioning and vitality and consists of 12 questions.
GDS | Within a week of the end of treatment (within 1 week of the completion of the 8-week treatment)
  This scale was developed by Yesavage et al. (1983). The Turkish adaptation of the scale was made by Ertan et al. The scale is self-reporting, aimed at the elderly, easy to answer and consists of 30 questions. A higher score indicates a higher level of depression.
Bioelectrical impedance analysis (BIA) | Within a week of the end of treatment (within 1 week of the completion of the 8-week treatment)
  Bioelectrical impedance analysis (BIA) measurement; It is a non-invasive measurement. It takes advantage of the different resistance of different tissues in the body to currents. A weak electric current is directed to the body and the impedance is measured. It is used to estimate body composition parameters such as total body water and fat-free mass.
Handgrip strength assessment | Within a week of the end of treatment (within 1 week of the completion of the 8-week treatment)
  During the assessment, the individual is seated upright on a chair without surface support for the arm being assessed. The arm to be measured is positioned in a free position, with the knee angle and elbow angle at 90 degrees. The subject is asked to squeeze the dynamometer with their fingers as hard and tight as possible. The measurements are repeated 3 times, with 10 seconds between them and each measurement being no less than 5 seconds, and any interventions that may affect the measurements during the assessment are avoided.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Erdoğan, Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All IPD collected